CLINICAL TRIAL: NCT00250354
Title: The Safety And Efficacy Of Risperidone Versus Placebo In Conduct Disorder In Mild, Moderate And Borderline Mentally Retarded Children Aged 5 To 12 Years
Brief Title: A Study of the Safety and Effectiveness of Risperidone for the Treatment of Conduct Disorder and Other Disruptive Behavior Disorders in Children Ages 5 to 12 With Mild, Moderate, or Borderline Mental Retardation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006007
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Conduct Disorder; Oppositional Defiant Disorder; Disruptive Behavior Disorder
Keywords: conduct disorder; oppositional deficit disorder; disruptive behavior disorder not otherwise specified; ADHD; risperidone; antipsychotropic agents; children
MeSH Terms: conditions — Conduct Disorder; Oppositional Defiant Disorder; Attention Deficit and Disruptive Behavior Disorders; Attention Deficit Disorder with Hyperactivity | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone oral solution

SUMMARY:
The purpose of the study is to assess the safety and effectiveness of oral risperidone (an antipsychotic medication) in the treatment of conduct disorder and other disruptive behavior disorders in children ages 5 to 12 with mild, moderate, or borderline mental retardation.

DETAILED DESCRIPTION:
Conduct and psychiatric disorders are found among a higher proportion of people with mental retardation than among people who are not mentally retarded. Among many different treatment approaches to conduct disorder are drug therapy, behavioral treatment, psychotherapy, cognitive and social learning. Studies have suggested that neuroleptic drugs, such as risperidone, may be beneficial in treating conduct disorder in mental retardation. This is a randomized, double-blind study to evaluate the effectiveness of risperidone compared with placebo in the treatment of children 5 to 12 years of age with mild, moderate, or borderline mental retardation who display destructive behaviors. The study has 2 phases: a run-in phase of 1 week and a treatment phase of 6 weeks. Patients receive placebo to be taken orally once a day during the first week (run-in). On the basis of scores on the Nisonger Child Behavior Rating Form (N-CBRF) after the first week, patients either continue in the double-blind treatment phase or discontinue the study. During the treatment phase patients receive risperidone oral solution once daily at a starting dose of 0.01 mg/kg body weight, increasing gradually at the investigator's discretion up to 0.06 mg/kg (maximum), or placebo for 6 weeks. A parent or caregiver evaluates the child's behavior and symptoms at scheduled office visits during the course of treatment. The primary measure of efficacy is the change from baseline to the end of treatment in the Conduct Problem subscale of the N-CBRF. Other efficacy assessments include the changes in the Aberrant Behavior Checklist (ABC), Behavioral Problems Inventory (BPI), and the Clinical Global Impression (CGI), a rating system used to evaluate the overall and severity of clinical change. Safety assessments include the incidence of adverse events throughout the study; weekly measurement of vital signs (pulse, temperature, blood pressure) and evaluation of the presence and severity of extrapyramidal symptoms by the Extrapyramidal Symptom Rating Scale (ESRS); and clinical laboratory tests (hematology, biochemistry, urinalysis) before study initiation and at end of treatment. The study hypothesis is that risperidone will be well tolerated and effective for the treatment of conduct disorder in children aged 5 to 12 years with mild, moderate, or borderline mental retardation. Risperidone oral solution 1.0 mg/mL once daily. Days 1 and 2 at a dose of 0.01 mg/kg body weight, Day 3 at a dose of 0.02 mg/kg, and increasing gradually up to 0.06 mg/kg (maximum) daily through 6 weeks. Dose may be increased or decreased at investigator's discretion

ELIGIBILITY:
Inclusion Criteria:

* Meets Axis I diagnosis criteria for Conduct Disorder or Oppositional Defiant Disorder or Disruptive Behavior Disorder not otherwise specified (DSM-IV, Diagnostic and Statistical Manual of Mental Diseases, 4th edition) and has a total rating of >=24 on the Nisonger Child Behavior Rating Form (N-CBRF) Conduct Problem Subscale. (Patients with conduct disorder who also meet DSM-IV criteria for Attention Deficit/Hyperactivity Disorder (AD/HD) are eligible.)
* meets DSM-IV Axis II diagnosis criteria for Mild Mental Retardation, Moderate Mental Retardation or Borderline Intellectual Functioning (diagnoses that represent intelligence quotients [IQs] ranging from 35 to 84)

Exclusion Criteria:

* DSM-IV diagnosis of Pervasive Development Disorder, Schizophrenia, or Other Psychotic Disorders
* head injury as cause of mental impairment
* seizure disorder currently requiring medication
* history of tardive dyskinesia (a condition of uncontrollable movements of the tongue, lips, face, trunk, hands and feet that is seen in patients receiving long-term medication with certain types of antipsychotic drugs) or neuroleptic malignant syndrome (a rare psychotropic-drug reaction, which may be characterized by confusion, reduced consciousness, high fever or pronounced muscle stiffness)
* known hypersensitivity, intolerance, or unresponsiveness to risperidone.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 1997-09; Study Completion 1999-08 (Actual)

PRIMARY OUTCOMES:
Change in the Conduct Problem subscale of the Nisonger Child Behavior Rating Form (N-CBRF) at end of treatment compared with baseline.

SECONDARY OUTCOMES:
Changes in Aberrant Behavior Checklist (ABC), Behavioral Problems Inventory (BPI), and Clinical Global Impression (CGI) at end of treatment compared with baseline; incidence of adverse events throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.

REFERENCES:
- [Result] Snyder R, Turgay A, Aman M, Binder C, Fisman S, Carroll A; Risperidone Conduct Study Group. Effects of risperidone on conduct and disruptive behavior disorders in children with subaverage IQs. J Am Acad Child Adolesc Psychiatry. 2002 Sep;41(9):1026-36. doi: 10.1097/00004583-200209000-00002. PMID 12218423